CLINICAL TRIAL: NCT01434498
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of GS-5885, GS-9451, Tegobuvir and Ribavirin; GS-5885, GS-9451 and Tegobuvir; GS-5885, GS-9451 and Ribavirin in Interferon Ineligible or Intolerant Subjects With Chronic Genotype 1a or 1b HCV Infection (Protocol No. GS US 248 0132)
Brief Title: GS-5885, GS-9451, Tegobuvir and Ribavirin (RBV) in Interferon Ineligible or Intolerant Subjects With Chronic Genotype 1a or 1b Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-248-0132
Record Dates: First submitted 2011-09-09; First posted 2011-09-15 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Genotype 1a or 1b HCV Infection
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Tegobuvir; Treatment naïve; HCV RNA; Polymerase inhibitor; Protease inhibitor; Interferon intolerant; Interferon ineligible; GS-9190; GS-9451; GS-5885
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir; GS-9451; tegobuvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): GS-5885, GS-9451, tegobuvir (GS-9190), and Copegus® for 24 weeks
  Interventions: Drug: GS-5885 tablet; Drug: GS-9451 tablet; Drug: tegobuvir capsule; Drug: ribavirin tablet
- Arm 2 (Active Comparator): GS-5885, GS-9451, tegobuvir (GS-9190), and a placebo matching ribavirin for 24 weeks
  Interventions: Drug: GS-5885 tablet; Drug: GS-9451 tablet; Drug: tegobuvir capsule; Drug: placebo matching ribavirin tablet
- Arm 3 (Active Comparator): GS-5885, GS-9451, a placebo matching tegobuvir, and Copegus® for 24 weeks
  Interventions: Drug: GS-5885 tablet; Drug: GS-9451 tablet; Drug: ribavirin tablet; Device: placebo matching tegobuvir capsule

INTERVENTIONS:
Drug: GS-5885 tablet — GS-5885 tablet, 90 mg, QD
Drug: GS-9451 tablet — GS-9451 tablet, 200 mg QD
Drug: tegobuvir capsule — tegobuvir capsule, 30 mg BID
  Arms: Arm 1; Arm 2
Drug: ribavirin tablet — ribavirin tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID)
  Arms: Arm 1; Arm 3
Drug: placebo matching ribavirin tablet — placebo matching ribavirin tablet, BID
  Arms: Arm 2
Device: placebo matching tegobuvir capsule — placebo matching tegobuvir capsule, BID
  Arms: Arm 3

SUMMARY:
This is a Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of GS-5885, GS-9451, Tegobuvir and Ribavirin; GS-5885, GS-9451 and Tegobuvir; GS-5885, GS-9451 and Ribavirin in Interferon Ineligible or Intolerant Subjects with Chronic Genotype 1a or 1b HCV Infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 and older with chronic HCV infection
* Liver biopsy results (performed no more than 3 years prior to Screening) indicating the absence of cirrhosis
* Monoinfection with HCV genotype 1a or 1b
* Interferon ineligible or intolerant
* Body mass index (BMI) between 18 and 40 kg/m2
* Use of highly effective contraception methods if female of childbearing potential or sexually active male
* Screening laboratory values within defined thresholds
* Has not been exposed to any investigational drug or device within 30 days of the Screening visit
* Able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

Exclusion Criteria:

* Prior treatment of HCV with any direct-acting antiviral (whether approved or experimental)
* Decompensated liver disease or cirrhosis
* Co-infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or another HCV genotype
* History of difficulty with blood collection and/or poor venous access
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non-HCV etiology
* Suspicion of hepatocellular carcinoma
* Clinically-relevant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Through 24 weeks of off-treatment follow-up
  To evaluate safety and tolerability of combination therapy with GS-5885, GS-9451, tegobuvir and ribavirin or GS-5885, GS-9451 and tegobuvir or GS-5885, GS-9451 and ribavirin. Safety will be assessed during the study through the reporting of adverse events, clinical laboratory tests, physical examinations, vital signs and 12-lead ECGs at various time points during the study.
Antiviral Activity | Through 24 weeks of off-treatment follow-up
  To evaluate antiviral efficacy as measured by sustained virologic response (defined as HCV RNA < lower limit of quantitation 24-weeks post-treatment) of combination therapy with GS-5885, GS-9451, tegobuvir and ribavirin or GS-5885, GS-9451 and tegobuvir or GS-5885, GS-9451 and ribavirin.

SECONDARY OUTCOMES:
Viral Dynamics | Through 10 days of therapy
  To characterize the viral dynamics of GS-5885, GS-9451 and tegobuvir. The median change from baseline in HCV RNA and time-weighted average change from baseline through Day 10 will be assessed based on plasma HCV RNA sampling times to characterize the viral dynamics of GS-5885, GS-9451 and tegobuvir.
Composite (or Profile) of Pharmacokinetics | predose, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
  To characterize the steady state pharmacokinetics of GS-5885, GS-9451, tegobuvir and ribavirin (if appropriate). Cmax, Tmax, Clast, Tlast, Ctau, λz, AUCtau and T ½

CONTACTS AND LOCATIONS:
Overall Officials: John McNally, PhD, Study Director — Gilead Sciences
Locations (49):
- United States (36):
  - California Liver Institute, Beverly Hills, California
  - SCTI Research Foundation Liver Center, Coronado, California
  - Scripps Clinic, La Jolla, California
  - University of California, San Diego, La Jolla, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Lightsource Medical, Los Angeles, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Center for Liver Diseases, Miami, Florida
  - Orlando Immunology Center (ACH), Orlando, Florida
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Saint Michael's Medical Center, Newark, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - The North Texas Research Institute, Arlington, Texas
  - The University of Texas Medical Branch, Galveston, Texas
  - The University of Texas Health Sciences Center at Houston, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Inova Fairfax Hospital Center for Liver Diseases, Falls Church, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (12):
  - University of Calgary, Calgary, Alberta
  - University Of Alberta Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - GIRI GI Research Institute, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hospital Saint-Luc DU CHUM, Montreal, Quebec
- Clinical Research Puerto Rico Inc, San Juan, Puerto Rico